CLINICAL TRIAL: NCT05301153
Title: Expression Levels of Interleukin 37 and Its Correlation With Autoantibodies and Disease Severity in Myasthenia Gravis Patients
Brief Title: Interleukin and Autoantibodies in Myasthenia Gravis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Radwa Medhat Ahmed El Galaly, Demonstrator at Medical Microbiology and Immunology Department, Assiut University
Other Study IDs: myasthenia1932022
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myasthenia Gravis cases: 1. Collection of Peripheral Blood Peripheral blood mononuclear cells (PBMCs) will be isolated from freshly drawn heparinized blood by ficoll density gradient centrifugation according to the manufacturer's protocol.
  2. Real-Time Reverse Transcription -PCR (RT-PCR) Real-time RT PCR will be performed on complementary DNA produced from 250 ng total RNA using the following primers Interleukin 37, F: 59-CAGTGAGGTCAGCGATTAGGAA-39 R: 59-TTAGTGAGCAGGTTTGGTGTTTT-39 b-actin, F: 59-CACCATTGGCAATGAGCGGTTC-39 R 59-AGGTCTTTGCGGATGTCCACGT-39.
  3. Autoantibodies detection:
  Detection of autoantibodies to muscle specific kinase (MuSK) and low-density lipoprotein receptor-related protein 4 (LRP4) serum levels by ELISA according to the manufacturer's protocol.
  Interventions: Diagnostic Test: real time PCR , ELISA
- Healthy Control: 1. Collection of Peripheral Blood Peripheral blood mononuclear cells (PBMCs) will be isolated from freshly drawn heparinized blood by ficoll density gradient centrifugation according to the manufacturer's protocol.
  2. Real-Time Reverse Transcription -PCR (RT-PCR) Real-time RT PCR will be performed on complementary DNA produced from 250 ng total RNA using the following primers Interleukin 37, F: 59-CAGTGAGGTCAGCGATTAGGAA-39 R: 59-TTAGTGAGCAGGTTTGGTGTTTT-39 b-actin, F: 59-CACCATTGGCAATGAGCGGTTC-39 R 59-AGGTCTTTGCGGATGTCCACGT-39.
  Interventions: Diagnostic Test: real time PCR , ELISA

INTERVENTIONS:
Diagnostic Test: real time PCR , ELISA — Real-time RT PCR will be performed on complementary DNA produced from 250 ng total RNA using the following primers Interleukin 37, F: 59-CAGTGAGGTCAGCGATTAGGAA-39 R: 59-TTAGTGAGCAGGTTTGGTGTTTT-39 b-actin, F: 59-CACCATTGGCAATGAGCGGTTC-39 R 59-AGGTCTTTGCGGATGTCCACGT-39. Detection of autoantibodies to muscle specific kinase (MuSK) and low-density lipoprotein receptor-related protein 4 (LRP4) serum levels by ELISA

SUMMARY:
Myasthenia gravis is a B-cell-mediated autoimmune disorders causing muscle weakness due to defective synaptic transmission at the neuromuscular junction caused by autoantibodies to acetylcholine receptors in (∼85%), muscle specific kinase in 6% and low-density lipoprotein receptor-related protein 4.The detection of these autoantibodies is very important not only in the diagnosis, but also for the stratification of Myasthenia Gravis patients into respective subgroups. These groups can differ in clinical manifestations, prognosis and response to therapies which become relevant for the development of antigen-specific therapies, targeting only the specific autoantibodies involved in the autoimmune response.

DETAILED DESCRIPTION:
Follicular T cells play a vital role during autoimmune disorders. The enhanced number or activation of these cells results in hyperproliferation of autoreactive B cells and overproduction of antibodies. Interleukin-37 is a newly identified immune-suppressive factor. It acts as an inhibitor of inflammation and plays an important regulatory role in both innate and adaptive immune responses. In Myasthenia Gravis, Cluster of differentiation 4+ T cell is the dominant cellular source for Interleukin-37 production directed to T follicular helper and B cells .It represses cell proliferation and secretion of autoantibody indicating that Interleukin-37 is a critical regulatory factor. The immunosuppressive features of Interleukin 37 contributing to autoimmune diseases are important and still poorly investigated. For this reason, the present study is designed to detect the level of expression of Interleukin 37 in Myasthenia Gravis patients and its correlation with autoantibodies serum levels and disease severity.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Diagnosis of Myasthenia Gravis.
2. Willingness to sample collection.

Exclusion Criteria:

1. History of chronic psychiatric or neurological disorder other than Myasthenia Gravis that can produce weakness or fatigue.
2. Severe systemic illness affecting life-expectancy ( chronic liver or kidney diseases).
3. History of autoimmune diseases, connective tissue diseases, , or genetic diseases.
4. Patients on large dosage of immune-suppressive treatment or Intravenous immunoglobulin in the recent 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The estimated minimum required sample size is 84 cases (42 case in each group). sample size was calculated using G*power software 3.1.9.7. As this study aims to detect the large difference between the the group of Myasthenia Gravis patients relative to the healthy controls, so the calculation based on determining the large effect size.
  Main statistical test is two tailed t-test to detect difference between two groups .
  Effect size = 0.8 Alpha = 0.05 Power = 0.95 Allocation ratio = 1
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Expression levels of Interleukin 37 | a year
  change in the expression levels of Interleukin 37 gene in the Myasthenia Gravis patients relative to the healthy control.

SECONDARY OUTCOMES:
Autoantibodies detection | a year
  Correlation of the gene expression levels with muscle specific kinase (MuSK) and low-density lipoprotein receptor-related protein (LRP4) autoantibodies serum level.

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Medhat, Dem, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fichtner ML, Jiang R, Bourke A, Nowak RJ, O'Connor KC. Autoimmune Pathology in Myasthenia Gravis Disease Subtypes Is Governed by Divergent Mechanisms of Immunopathology. Front Immunol. 2020 May 27;11:776. doi: 10.3389/fimmu.2020.00776. eCollection 2020. PMID 32547535
- [Result] Lazaridis K, Tzartos SJ. Autoantibody Specificities in Myasthenia Gravis; Implications for Improved Diagnostics and Therapeutics. Front Immunol. 2020 Feb 14;11:212. doi: 10.3389/fimmu.2020.00212. eCollection 2020. PMID 32117321
- [Result] Crotty S. Follicular helper CD4 T cells (TFH). Annu Rev Immunol. 2011;29:621-63. doi: 10.1146/annurev-immunol-031210-101400. PMID 21314428
- [Result] King C, Tangye SG, Mackay CR. T follicular helper (TFH) cells in normal and dysregulated immune responses. Annu Rev Immunol. 2008;26:741-66. doi: 10.1146/annurev.immunol.26.021607.090344. PMID 18173374
- [Result] Liu Z, Zhu L, Lu Z, Chen H, Fan L, Xue Q, Shi J, Li M, Li H, Gong J, Shi J, Wang T, Jiang ML, Cao R, Meng H, Wang C, Xu Y, Zhang CJ. IL-37 Represses the Autoimmunity in Myasthenia Gravis via Directly Targeting Follicular Th and B Cells. J Immunol. 2020 Apr 1;204(7):1736-1745. doi: 10.4049/jimmunol.1901176. Epub 2020 Feb 28. PMID 32111731